CLINICAL TRIAL: NCT04379336
Title: Reducing Morbidity and Mortality in Health Care Workers Exposed to SARS-CoV-2 by Enhancing Non-specific Immune Responses Through Bacillus Calmette-Guérin Vaccination, a Randomized Controlled Trial
Brief Title: BCG Vaccination for Healthcare Workers in COVID-19 Pandemic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TASK Applied Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TASK-008 BCG-CORONA
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Sars-CoV2
Keywords: Blinded; Randomized controlled; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Efficacy will be determined based on documented SARS-CoV-2 infection and incidence of hospitalization. The analysis will be an intention-to-treat analysis with estimation of hazard ratio between the two arms using a Cox proportional hazard model. Adverse events will be summarized using descriptive statistics per study arm. The analysis will be a model-based analysis of cumulative data on general health status as a function of risk factors, treatment arm and time.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacille Calmette-Guérin (BCG) (Experimental): Participants will receive an intradermal injection of 0.1ml of the suspended BCG vaccine which accounts for 0.075mg of attenuated Mycobacterium bovis. BCG-Vaccin SSI [Statens Serum Institut], Danish strain 1331.
  Interventions: Biological: Bacille Calmette-Guérin (BCG)
- Placebo (Placebo Comparator): The placebo used for this study is 0.9% Sodium Chloride (NaCl). Participants that are randomized to the control arm will receive a placebo injection of 0.1ml 0.9% NaCl, which is the same volume and has the same colour as the suspended BCG vaccine.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: Bacille Calmette-Guérin (BCG) — BCG vaccine will be given intradermally in the upper arm after randomization.
  Other Names: BCG-Vaccin SSI [Statens Serum Institut], Danish strain 1331
  Arms: Bacille Calmette-Guérin (BCG)
Other: Placebo Comparator — Placebo injection will be given intradermally in the upper arm after randomization.
  Other Names: 0.9% Sodium Chloride
  Arms: Placebo

SUMMARY:
A novel betacoronavirus, SARS-CoV-2, is spreading rapidly throughout the world. A large epidemic in South Africa may overwhelm available hospital capacity and healthcare resources which would be worsened by absenteeism of healthcare workers and other frontline staff (HCW). Strategies to prevent morbidity and mortality of HCW are desperately needed to safeguard continuous patient care. Bacillus Calmette-Guérin (BCG) is a vaccine against tuberculosis (TB), with protective non-specific effects against other respiratory tract infections in in vitro and in vivo studies, with reported morbidity and mortality reductions as high as 70%. We hypothesize that a BCG vaccination may reduce the morbidity and mortality of healthcare workers during the COVID-19 outbreak in South Africa.

DETAILED DESCRIPTION:
Morbidity and mortality attributable to COVID-19 is devastating global health systems and economies. Bacillus Calmette Guérin (BCG) vaccination has been in use for many decades to prevent severe forms of tuberculosis in children. Studies have also shown a combination of improved long-term innate or trained immunity (through epigenetic reprogramming of myeloid cells) and adaptive responses after BCG vaccination, which leads to non-specific protective effects in adults. Observational studies have shown that countries with routine BCG vaccination programs have significantly less reported cases and deaths of COVID-19, but such studies are prone to significant bias and need confirmation. To date, in the absence of direct evidence, WHO does not recommend BCG for the prevention of COVID-19.

This project aims to investigate in a timely manner whether and why BCG-revaccination can reduce infection rate and/or disease severity in health care workers during the SARS-CoV-2 outbreak in South Africa. These objectives will be achieved with a blinded, randomised controlled trial of BCG revaccination versus placebo in exposed front-line staff in hospitals in Cape Town. Observations will include the rate of infection with COVID-19 as well as the occurrence of mild, moderate or severe ambulatory respiratory tract infections, hospitalisation, need for oxygen, mechanical ventilation or death. HIV-positive individuals will be excluded. Safety of the vaccines will be monitored. A secondary endpoint is the occurrence of latent or active tuberculosis. Initial sample size and follow-up duration is at least 500 workers and 52 weeks. Statistical analysis will be model-based and ongoing in real time with frequent interim analyses and optional increases of both sample size or observation time, based on the unforeseeable trajectory of the South African COVID-19 epidemic, available funds and recommendations of an independent data and safety monitoring board.

Given the immediate threat of the SARS-CoV-2 epidemic the trial has been designed as a pragmatic study with highly feasible endpoints that can be continuously measured. This allows for the most rapid identification of a beneficial outcome that would lead to immediate dissemination of the results, vaccination of the control group and outreach to the health authorities to consider BCG vaccination for all qualifying health care workers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years
* HCW or other frontline staff currently in contact with, or anticipated to be in contact with, patients with SARS-CoV-2 infection.
* Ability and willingness to provide informed consent.
* Can be reached by mobile phone for follow-up

Exclusion Criteria:

* Known allergy to (components of) the BCG vaccine or serious reaction to prior BCG administration.
* Known active tuberculosis or any other active or uncontrolled condition that, in the opinion of the investigator or designee, makes participation unsafe or makes it difficult to collect follow-up data over the study period.
* HIV-1 infection

  - NOTE: If evidence of recent HIV negative test is not available, rapid point-of-care testing will be undertaken as part of screening with a separate informed consent process.
* Symptoms of respiratory tract infection which, in the opinion of the investigator or designee, is likely to interfere with the objectives of the study.
* Known medical history of any of the following immunocompromised states:

  * Neutropenia (less than 500 neutrophils/mm3)
  * Lymphopenia (less than 400 lymphocytes/mm3)
  * Solid organ or bone marrow transplantation
  * Primary immunodeficiency
  * Active solid or non-solid malignancy or lymphoma within the prior two years
  * Pregnancy and breastfeeding
* Current treatment with the following medications:

  * Chemotherapy
  * Anti-cytokine therapies
  * Current treatment with oral or intravenous steroids defined as daily doses of 10mg prednisone or equivalent for longer than 3 months
  * Any experimental, unproven treatment against SARS-CoV-2 infection or COVID-19 including but not limited to chloroquine, hydroxychloroquine, remdesivir, lopinavir/ritonavir and interferon beta-1a.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Incidence of HCWs hospitalized due to COVID-19 per arm | 52 weeks
  To compare the incidence of HCWs hospitalized due to COVID-19 per arm.

SECONDARY OUTCOMES:
Incidence of SARS-CoV-2 infection per arm | 52 weeks
  To determine the incidence of SARS-CoV-2 infection in HCW by molecular or serological testing (as available) at entry, 10, 26 and/or 52 weeks.
Incidence of upper respiratory tract infections per arm | 52 weeks
  To compare the incidence of symptoms of upper respiratory tract infection per arm.
Days of unplanned absenteeism due to COVID-19 or any reason per arm | 52 weeks
  To compare the number of days of (unplanned) absenteeism because of documented SARS-CoV-2 infection, COVID-19 or any reason per arm.
Incidence of hospitalization for any reason per arm | 52 weeks
  To compare the incidence of hospitalization of HCW for any reason per arm.
Incidence of intensive care unit admission per arm | 52 weeks
  To compare the incidence of intensive care admission of HCW due to COVID-19 or any reason per arm.
Incidence of death per arm | 52 weeks
  To compare the incidence of death of HCW due to COVID-19 or any reason per arm.
Prevalence of latent TB infection | 52 weeks
  To describe the prevalence of latent TB infection as determined by interferon gamma release assay (IGRA) at enrolment and at week 52.
Incidence of active TB per arm | 52 weeks
  To compare the incidence of active TB of HCW per arm.
Compare the effect of latent TB on morbidity and mortality due to COVID-19 per arm | 52 weeks
  To compare the effect of latent TB infection on morbidity and mortality of HCW due to COVID-19 per arm. The risk of morbidity and mortality of latent TB infected individuals is not known, we will examine whether there is a higher risk of disease severity and poor outcomes in this group.
Incidence of treatment related adverse events | 52 weeks
  To compare the incidence of grade 2 or higher adverse events and vaccination site reactions per arm.

CONTACTS AND LOCATIONS:
Locations (1):
- TASK Foundation, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared among researchers included in the protocol team at this stage.

REFERENCES:
- [Background] Netea MG, Schlitzer A, Placek K, Joosten LAB, Schultze JL. Innate and Adaptive Immune Memory: an Evolutionary Continuum in the Host's Response to Pathogens. Cell Host Microbe. 2019 Jan 9;25(1):13-26. doi: 10.1016/j.chom.2018.12.006. PMID 30629914
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Joosten LA, Ifrim DC, Saeed S, Jacobs C, van Loenhout J, de Jong D, Stunnenberg HG, Xavier RJ, van der Meer JW, van Crevel R, Netea MG. Bacille Calmette-Guerin induces NOD2-dependent nonspecific protection from reinfection via epigenetic reprogramming of monocytes. Proc Natl Acad Sci U S A. 2012 Oct 23;109(43):17537-42. doi: 10.1073/pnas.1202870109. Epub 2012 Sep 17. PMID 22988082
- [Derived] van Wijk RC, Mockeliunas L, Upton CM, Peter J, Diacon AH, Simonsson USH. Seasonal influence on respiratory tract infection severity including COVID-19 quantified through Markov Chain modeling. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1250-1261. doi: 10.1002/psp4.13006. Epub 2023 Jul 10. PMID 37401774
- [Derived] Upton CM, van Wijk RC, Mockeliunas L, Simonsson USH, McHarry K, van den Hoogen G, Muller C, von Delft A, van der Westhuizen HM, van Crevel R, Walzl G, Baptista PM, Peter J, Diacon AH; BCG CORONA Consortium. Safety and efficacy of BCG re-vaccination in relation to COVID-19 morbidity in healthcare workers: A double-blind, randomised, controlled, phase 3 trial. EClinicalMedicine. 2022 Jun;48:101414. doi: 10.1016/j.eclinm.2022.101414. Epub 2022 May 12. PMID 35582122